CLINICAL TRIAL: NCT04006912
Title: The Influence of Different Preoperative Decision Schemes on the Visual Quality After Toric Intraocular Lens Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuwen2019-079
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2020-12

CONDITIONS: Recruitment of Participants
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal residual theoretical astigmatism group (Experimental)
  Interventions: Procedure: phacoemulsification and Toric intraocular lens implantation
- Steep meridian incision design group (Active Comparator)
  Interventions: Procedure: phacoemulsification and Toric intraocular lens implantation

INTERVENTIONS:
Procedure: phacoemulsification and Toric intraocular lens implantation — A clear corneal incision is made in a different position

SUMMARY:
To study the Influence of Different Preoperative Decision Schemes on the Visual Quality After Toric Intraocular Lens Implantation

ELIGIBILITY:
Inclusion Criteria:

1. Age-related cataract (age 55-80)
2. Corneal astigmatism is greater than 1.0D
3. Patients who are willing to implant Toric IOL

Exclusion Criteria:

1. Previous or present eye diseases, such as glaucoma, eye trauma, etc
2. High refractive error
3. Previous eye surgery
4. Irregular astigmatism of the cornea

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Actual residual astigmatism after surgery | 1 week postoperation
  The actual residual astigmatism value after the operation is measured with the phoropter
Actual residual astigmatism after surgery | 1 month postoperation
  The actual residual astigmatism value after the operation is measured with the phoropter
Actual residual astigmatism after surgery | 3 month postoperation
  The actual residual astigmatism value after the operation is measured with the phoropter

SECONDARY OUTCOMES:
uncorrected distance visual acuity (UDVA) | 1 week postoperation
  uncorrected distance visual acuity (UDVA) is observed in each group
uncorrected distance visual acuity (UDVA) | 1 month postoperation
  uncorrected distance visual acuity (UDVA) is observed in each group
uncorrected distance visual acuity (UDVA) | 3 month postoperation
  uncorrected distance visual acuity (UDVA) is observed in each group
Theoretical residual astigmatism after surgery | 1 week postoperation
  The theoretical residual astigmatism is obtained by TECNIS Toric online calculator
Theoretical residual astigmatism after surgery | 1 month postoperation
  The theoretical residual astigmatism is obtained by TECNIS Toric online calculator
Theoretical residual astigmatism after surgery | 3 month postoperation
  The theoretical residual astigmatism is obtained by TECNIS Toric online calculator
Postoperative Totic intraocular lens rotation angle | 1 week postoperation
  Postoperative Totic intraocular lens rotation angle is observed in each group
Postoperative Totic intraocular lens rotation angle | 1 month postoperation
  Postoperative Totic intraocular lens rotation angle is observed in each group
Postoperative Totic intraocular lens rotation angle | 3 month postoperation
  Postoperative Totic intraocular lens rotation angle is observed in each group
Postoperative astigmatism and astigmatism axial of cornea | 1 week postoperation
  Postoperative astigmatism and astigmatism axial of cornea are measured with Pentacam
Postoperative astigmatism and astigmatism axial of cornea | 1 month postoperation
  Postoperative astigmatism and astigmatism axial of cornea are measured with Pentacam
Postoperative astigmatism and astigmatism axial of cornea | 3 month postoperation
  Postoperative astigmatism and astigmatism axial of cornea are measured with Pentacam
Corneal Aberrations | 1 week postoperation
  Corneal aberrations are measured with OPD-Scan Ⅲ
Corneal Aberrations | 1 month postoperation
  Corneal aberrations are measured with OPD-Scan Ⅲ
Corneal Aberrations | 3 month postoperation
  Corneal aberrations are measured with OPD-Scan Ⅲ

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Yu X, Wang J, Lin X, Xu D, Ni S, Sheng S, Xu W. Effect of two different preoperative calculation schemes on visual outcomes of patients after toric intraocular lens implantation. Int Ophthalmol. 2023 Feb;43(2):491-501. doi: 10.1007/s10792-022-02447-7. Epub 2022 Aug 6. PMID 35932419